CLINICAL TRIAL: NCT02822755
Title: Effectiveness of Individualized Video Recordings Versus Conventional Printed Instructions on Home Exercise Program Adherence in Physical Therapy
Brief Title: Home Exercise Adherence in Physical Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data collection sites lost research personnel that were recruiting subjects.
Sponsor: Evan J. Petersen (Other)
Responsible Party: Sponsor-Investigator, Evan J. Petersen, Dr., PT, DSc, OCS, FAAOMPT, University of the Incarnate Word
Organization: University of the Incarnate Word (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UniversityIW
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Adherence
Keywords: Exercise; Adherence; Physical Therapy
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Video Recording Group (Experimental): The experimental group participants will be recorded on their personal smartphone performing their prescribed exercises with individualized instruction from the participating physical therapist. The prescribing therapist will record participants on their own smartphones doing the exercise program in the clinic so that participants can have that video recording of the exercises to help remind them how to do the exercises properly at home. Participants will not be asked to record themselves performing future exercise sessions as documentation of improvement. Intervention: Home Exercise Program and Adherence Logs
  Interventions: Other: Home Exercise Program and Adherence Logs
- Conventional Printed Group (Active Comparator): The active comparator group will receive individualized instruction from the participating physical therapist on how to perform their home exercise program as well as printed instructions of the exercises. No video recording of the control group participants will be performed. Intervention: Home Exercise Program and Adherence Logs
  Interventions: Other: Home Exercise Program and Adherence Logs

INTERVENTIONS:
Other: Home Exercise Program and Adherence Logs — Both groups will receive physical therapy prescribed home exercises and be asked to record adherence to their program on an exercise log.
  Other Names: HEP

SUMMARY:
The purpose of this study is to determine the effectiveness of an individualized video recording in improving adherence in home exercise programs for orthopaedic physical therapy patients.

Specific aims:

1. Evaluate whether individualized video recordings improve adherence with home exercise programs (HEP) as compared with conventional printed instructions measured by a self-report exercise log. (1-tail analysis)

DETAILED DESCRIPTION:
This investigation will focus on the specific issues surrounding adherence to the use of individualized video recordings via smartphone versus conventional printed instructions in patients with orthopaedic injuries. The data reported will be used to explore the feasibility and potential benefits of smartphone usage for home exercise adherence.

ELIGIBILITY:
Inclusion Criteria:

* Participants who can read and understand the English language,
* adults between 18-65 years of age,
* have a referral to an outpatient physical therapy clinic for an orthopaedic condition, and
* who own a smartphone with video recording capabilities and available data storage space (at least 500 MB or 0.5 GB).

Exclusion Criteria:

* Individuals referred for non-orthopaedic conditions,
* individuals currently on an established, prescribed home exercise program,
* individuals requiring more than 4 home exercises at one time as part of their rehabilitation program, and
* individuals who do not own a smartphone device with the required storage and recording specifications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Home Exercise Adherence | Weekly for 6 weeks
  Data will be recorded via a self-reported exercise log that includes number of days exercises were completed per week. Participants will record the number of days participants did "All" of the program (defined as doing 100% of their exercises), "Most" of the program (defined as doing 75% of their exercises), "Some" of the program (defined as doing 50% of their program, and "None" of the program (defined as doing 0% of their exercise program).

CONTACTS AND LOCATIONS:
Overall Officials: Evan J Petersen, PT, DSc, Study Chair — University of the Incarnate Word
Locations (1):
- Texas Physical Therapy Specialists, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
All individual data will be reported as a group

REFERENCES:
- [Background] Gonzalez JS, McCarl LA, Wexler D DD, Cagliero E, Delahanty L, Soper TD, Goldman V, Knauz R, Safren SA. Cognitive Behavioral Therapy for Adherence and Depression (CBT-AD) in Type 2 Diabetes. J Cogn Psychother. 2010 Nov 1;24(4):329-343. doi: 10.1891/0889-8391.24.4.329. PMID 23667294
- [Background] Hammer C, Degerfeldt L, Denison E. Mechanical diagnosis and therapy in back pain: Compliance and social cognitive theory. Adv Physiother. 2007;9(4):190-197.
- [Background] Marks R, Allegrante JP. Chronic osteoarthritis and adherence to exercise: a review of the literature. J Aging Phys Act. 2005 Oct;13(4):434-60. doi: 10.1123/japa.13.4.434. PMID 16301755
- [Background] Papaioannou A, Kennedy CC, Dolovich L, Lau E, Adachi JD. Patient adherence to osteoporosis medications: problems, consequences and management strategies. Drugs Aging. 2007;24(1):37-55. doi: 10.2165/00002512-200724010-00003. PMID 17233546
- [Background] Conraads VM, Deaton C, Piotrowicz E, Santaularia N, Tierney S, Piepoli MF, Pieske B, Schmid JP, Dickstein K, Ponikowski PP, Jaarsma T. Adherence of heart failure patients to exercise: barriers and possible solutions: a position statement of the Study Group on Exercise Training in Heart Failure of the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2012 May;14(5):451-8. doi: 10.1093/eurjhf/hfs048. Epub 2012 Apr 11. PMID 22499542
- [Background] Jordan JL, Holden MA, Mason EE, Foster NE. Interventions to improve adherence to exercise for chronic musculoskeletal pain in adults. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD005956. doi: 10.1002/14651858.CD005956.pub2. PMID 20091582
- [Background] Yuen HK, Wang E, Holthaus K, Vogtle LK, Sword D, Breland HL, Kamen DL. Self-reported versus objectively assessed exercise adherence. Am J Occup Ther. 2013 Jul-Aug;67(4):484-9. doi: 10.5014/ajot.2013.007575. PMID 23791324
- [Background] Holden MA, Haywood KL, Potia TA, Gee M, McLean S. Recommendations for exercise adherence measures in musculoskeletal settings: a systematic review and consensus meeting (protocol). Syst Rev. 2014 Feb 10;3:10. doi: 10.1186/2046-4053-3-10. PMID 24512976
- [Background] Kramer A, Dettmers C, Gruber M. Exergaming with additional postural demands improves balance and gait in patients with multiple sclerosis as much as conventional balance training and leads to high adherence to home-based balance training. Arch Phys Med Rehabil. 2014 Oct;95(10):1803-9. doi: 10.1016/j.apmr.2014.04.020. Epub 2014 May 10. PMID 24823959
- [Background] Friedrich M, Cermak T, Maderbacher P. The effect of brochure use versus therapist teaching on patients performing therapeutic exercise and on changes in impairment status. Phys Ther. 1996 Oct;76(10):1082-8. doi: 10.1093/ptj/76.10.1082. PMID 8863761
- [Background] Harkapaa K, Jarvikoski A, Mellin G, Hurri H. A controlled study on the outcome of inpatient and outpatient treatment of low back pain. Part I. Pain, disability, compliance, and reported treatment benefits three months after treatment. Scand J Rehabil Med. 1989;21(2):81-9. PMID 2526364
- [Background] Khalil H, Quinn L, van Deursen R, Martin R, Rosser A, Busse M. Adherence to use of a home-based exercise DVD in people with Huntington disease: participants' perspectives. Phys Ther. 2012 Jan;92(1):69-82. doi: 10.2522/ptj.20100438. Epub 2011 Sep 29. PMID 21960468
- [Background] Roddey TS, Olson SL, Gartsman GM, Hanten WP, Cook KF. A randomized controlled trial comparing 2 instructional approaches to home exercise instruction following arthroscopic full-thickness rotator cuff repair surgery. J Orthop Sports Phys Ther. 2002 Nov;32(11):548-59. doi: 10.2519/jospt.2002.32.11.548. PMID 12449254